CLINICAL TRIAL: NCT04533672
Title: Multiparametric Magnetic Resonance Imaging (MRI) to Improve Bladder Cancer Staging and Treatment Decision-making
Acronym: SBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SBCT
Record Dates: First submitted 2020-08-23; First posted 2020-08-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single study arm (Experimental)
  Interventions: Diagnostic Test: MRI Sequences

INTERVENTIONS:
Diagnostic Test: MRI Sequences — New multiparametric MRI techniques

SUMMARY:
The therapeutic approach to bladder cancer is strongly dependent on tumor stage and grade. Patients with non-muscle-invasive tumors (NMIBC) are usually treated with surgical resection of the tumor alone, whereas patients with muscle-invasive tumors (MIBC) ideally undergo neoadjuvant chemotherapy (NCT) and subsequent cystectomy. Magnetic Resonance Imaging (MRI) is emerging as a new staging modality, given its non-invasiveness and excellent soft tissue contrast. However, more advanced multiparametric MRI techniques are yet to be comprehensively investigated in patients with bladder cancer. Recently, genetic characteristics of bladder tumors have been identified that show significant impact on response rates to neoadjuvant treatment. The combination of new multiparametric MRI (mpMRI) techniques and genetic analyses of the tumor might allow for a better assessment of the expected clinical course of the disease and support more personalized treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed or suspected primary bladder cancer and a circumscribed tumor/focal thickening of the bladder wall on initial imaging (ultrasound, CT) or cystoscopy with an approx. size of ≥ 1.5 cm/for which at least 2-3 TUR-B resection loops are necessary
* Informed consent as documented by signature (Informed Consent Form)

Exclusion Criteria:

* Prior TUR-B or other bladder treatment, prior treated bladder cancers, prior pelvic irradiation
* Women who are pregnant or breast-feeding. Female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of childbearing potential.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Patients with non-MRI compatible metallic or electronic implants, devices or metallic foreign bodies (cardiac pacemaker, shrapnel, cochlea implants, neurostimulator, or other non-MRI compatible implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Muscle-invasiveness | through study completion, an average of 4 years
  Presence of tumor infiltration into the muscular bladder wall, as per pathology report (infiltration: yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No